CLINICAL TRIAL: NCT04339907
Title: Uncovering Inflammatory Mediators of Glaucoma Pathogenesis After Corneal Transplantation in Aqueous Humor and Tears
Brief Title: Inflammatory Mediators of Glaucoma After Corneal Transplantation (AH-Tears)
Acronym: AH-Tears
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 20.004
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Glaucoma; Corneal Transplantation; Inflammation
Keywords: Boston keratoprosthesis type 1; Glaucoma; Aqueous Humor; Tears; Inflammation; Penetrating keratoplasty
MeSH Terms: conditions — Glaucoma; Inflammation; Lacerations

STUDY DESIGN:
Intervention Model Description: 5 groups will be compared:
  * participant needing cataract surgery without glaucoma
  * participant needing glaucoma filtration surgery without prior corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis)
  * participant needing corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis), with or without glaucoma
  * participant needing intraocular surgery (cataract, retina or glaucoma) with prior corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis)
  * participant needing glaucoma filtration surgery with prior corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cataract surgery only (Sham Comparator): Participants needing cataract surgery, without glaucoma or any other corneal diseases.
  Interventions: Other: Sampling of tears; Other: Sampling of aqueous humor
- Glaucoma surgery only (Sham Comparator): Participants needing glaucoma filtration surgery, without any prior corneal transplantation.
  Interventions: Other: Sampling of tears; Other: Sampling of aqueous humor
- Corneal transplantation (Experimental): Participants needing corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis), with or without glaucoma.
  This allows analyzing samples at baseline (time 0), at the time of the corneal transplantation procedure.
  Interventions: Other: Sampling of tears; Other: Sampling of aqueous humor
- Intraocular surgery following corneal transplantation (Experimental): Participants needing intraocular surgery (cataract, retina or glaucoma), with prior corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis).
  This allows analyzing samples during the potential development or progression of glaucoma in participants who have previously undergone corneal transplantation.
  Interventions: Other: Sampling of tears; Other: Sampling of aqueous humor
- Glaucoma surgery following corneal transplantation (Experimental): Participants needing glaucoma filtration surgery, with prior corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis).
  This allows analyzing samples once glaucoma is confirmed in participants who have previously undergone corneal transplantation.
  Interventions: Other: Sampling of tears; Other: Sampling of aqueous humor

INTERVENTIONS:
Other: Sampling of tears — Tears will be collected at the start of any of surgery for which the participant presents. It will be collected using a tear-wash method to allow for protein collection. 0.06 ml of saline solution 0.9% will be instilled on the ocular surface. The participants will turn their eyes with eyes closed. The tear-wash fluid will be collected from the inferior fornix of the eye using a micropipette. Tear-was fluid will be placed in codified tubes stored at -150 degrees.
Other: Sampling of aqueous humor — Aqueous humor will be collected at the start of any of surgery for which the participant presents. A paracentesis of the anterior chamber is a common first step in intraocular surgeries. Aqueous humor is then commonly diluted with viscoelastic material injected inside the anterior chamber to avoid collapse of the anterior chamber. This way, the aqueous humor is commonly diluted or replaced entirely by the viscoelastic material injected during intraocular surgeries. A volume of 0.1 ml of aqueous humor will be taken by paracentesis using a 30-gauge needle connected to a 1-ml syringe. It consists of less than half of the total volume of aqueous humor in the eye. Aqueous humor will be placed in codified tubes stored at -80 degrees.

SUMMARY:
Glaucoma is the most common threat to vision rehabilitation in patients with Boston keratoprosthesis type 1 (KPro) implantation. High intraocular pressure (IOP) is the most important risk factor for glaucoma and may lead to irreversible retinal and optic nerve damage. Glaucoma drainage device (GDD) surgery is used to divert aqueous humor (AH) from the anterior chamber to an external reservoir to regulate flow and decrease the IOP. The AH is in direct communication with any corneal damage or surgery undertaken in the anterior chamber and can serve as a source of potential biomarkers to detect early inflammatory or glaucomatous changes. Tears are also one of the most accessible and non-invasive source of biomarkers, especially in Kpro eyes where the central optic allows communication between aqueous humor and the tears at the surface of the eye. The investigators propose to test the hypothesis that distinct inflammatory mediators in the AH and tears can serve as biomarkers for glaucoma development and progression after CT, making them specifically amenable to targeted treatment strategies to minimize vision loss.

DETAILED DESCRIPTION:
The only curative treatment for corneal diseases that progress to vision loss is corneal transplantation (CT). Penetrating keratoplasty (PK) involves the surgical replacement of the host cornea with a donor cornea. In cases of graft failure with standard PK, the Boston keratoprosthesis (KPro), the most common artificial cornea, can alternatively restore vision rapidly. A current limitation in the use of KPro is that the vast majority of patients are at high risk of developing glaucoma. Glaucoma contributes to significant ocular morbidity after CT surgery and is the leading cause of irreversible vision loss after CT. High intraocular pressure (IOP) is the most important risk factor for glaucoma and may lead to irreversible retinal and optic nerve damage. Glaucoma is treated using drops or surgery to reduce IOP. When IOP-lowering drugs and laser surgery fail, glaucoma drainage device (GDD) surgery is used to divert aqueous humor (AH) from the anterior chamber to an external reservoir to regulate flow and decrease the IOP. The cause and mechanisms of glaucoma development and progression following CT are still unknown. Neuroinflammation has been suggested to play a key role in glaucomatous damage following CT. The role of inflammatory biomarkers in glaucoma pathogenesis after CT remains poorly understood and must be further studied. The AH is in direct communication with any corneal damage or surgery undertaken in the anterior chamber and can serve as a source of potential biomarkers to detect inflammatory changes in glaucoma. Tears are also one of the most accessible and non-invasive source of biomarkers, especially in Kpro eyes where the central optic allows communication between AH and the tears at the surface of the eye. Full thickness corneal transplantation (penetrating keratoplasty and Boston KPro) and intraocular surgeries for glaucoma, cataract and retina that are required by the participants of the study offer the opportunity to have access to the AH and tears in an accessible and safe way, without additional risks. These samples of AH and tears will be analyzed for multiple inflammatory mediators simultaneously.

HYPOTHESIS:

The investigators propose to test the hypothesis that distinct inflammatory mediators in the AH and tears can serve as biomarkers for glaucoma development and progression after CT, making them specifically amenable to targeted treatment strategies to minimize vision loss.

OBJECTIVES:

1. To examine the (a) presence and (b) concentration of inflammatory mediators in glaucoma after corneal transplantation.
2. To examine the correlation between the presence and concentration of inflammatory mediators and clinical ophthalmological data.
3. To examine the correlation between the inflammatory mediators found in aqueous humor and tears.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or older
* Informed consent
* Ability to be followed for the duration of the study
* Presence of ocular disease specified for each group

Specific criteria for each group:

* Group 1 : have no glaucoma and no systemic diseases
* Group 2 : need to have glaucoma filtration surgery without prior corneal transplantation
* Group 3 : need to have corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis), with or without glaucoma
* Group 4 : need to have intraocular surgery after prior corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis)
* Group 5 : need to have glaucoma filtration surgery with prior corneal transplantation (penetrating keratoplasty or Boston keratoprosthesis)

Exclusion Criteria:

* Aged less than 18
* Inability to give informed consent
* Presence of ocular diseases other than those studied herein

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Concentration of inflammatory mediators in aqueous humor | Baseline
  Concentration (pg/mL) of inflammatory mediators in aqueous humor measured by ELISA multiplex.
Concentration of inflammatory mediators in tears | Baseline
  Concentration (pg/mL) of inflammatory mediators in tears measured by ELISA multiplex.
Correlation between tears and aqueous humor | Baseline
  Correlation between the concentration of inflammatory mediators in tears and aqueous humor, determined by Spearman correlation test.

SECONDARY OUTCOMES:
Incidence of anterior structural changes | Baseline, 3 months, 6 months, 12 months
  Incidence of anterior structural changes in the eye (iris, iridocorneal angle, trabecular meshwork, cornea), evaluated by anterior segment optical coherence tomography (AS-OCT) imaging.
Change of visual acuity through time | Baseline, 3 months, 6 months, 12 months
  Change of visual acuity at each time point compared to baseline visual acuity. The visual acuity is measured using the Snellen chart.
Proportion of participants with visual field loss of 30% or more | Baseline, 3 months, 6 months, 12 months
  Proportion of participants with visual field loss of 30% or more at each time point, measured using the automated Humphrey 24-2 visual field. The loss of 30% or more of visual field is calculated using the baseline test as reference.
Intraocular pressure | Baseline, 3 months, 6 months, 12 months
  Evaluation of intraocular pressure (units of mmHg) at each time point using Goldman tonometry.
Incidence of posterior structural changes | Baseline, 3 months, 6 months, 12 months
  Incidence of posterior structural changes in the eye (optic nerve and retina), evaluated by spectral domain optical coherence tomography (SD-OCT) imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Younes Agoumi, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Mona Harissi-Dagher, MD, Study Director — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szigiato AA, Bostan C, Nayman T, Harissi-Dagher M. Long-term visual outcomes of the Boston type I keratoprosthesis in Canada. Br J Ophthalmol. 2020 Nov;104(11):1601-1607. doi: 10.1136/bjophthalmol-2019-315345. Epub 2020 Feb 17. PMID 32066560
- [Background] Wang Q, Harissi-Dagher M. Characteristics and management of patients with Boston type 1 keratoprosthesis explantation--the University of Montreal Hospital Center experience. Am J Ophthalmol. 2014 Dec;158(6):1297-1304.e1. doi: 10.1016/j.ajo.2014.08.037. Epub 2014 Aug 28. PMID 25174898
- [Background] Crnej A, Paschalis EI, Salvador-Culla B, Tauber A, Drnovsek-Olup B, Shen LQ, Dohlman CH. Glaucoma progression and role of glaucoma surgery in patients with Boston keratoprosthesis. Cornea. 2014 Apr;33(4):349-54. doi: 10.1097/ICO.0000000000000067. PMID 24531120
- [Background] Aldave AJ, Kamal KM, Vo RC, Yu F. The Boston type I keratoprosthesis: improving outcomes and expanding indications. Ophthalmology. 2009 Apr;116(4):640-51. doi: 10.1016/j.ophtha.2008.12.058. Epub 2009 Feb 25. PMID 19243830
- [Background] Baltaziak M, Chew HF, Podbielski DW, Ahmed IIK. Glaucoma after corneal replacement. Surv Ophthalmol. 2018 Mar-Apr;63(2):135-148. doi: 10.1016/j.survophthal.2017.09.003. Epub 2017 Sep 18. PMID 28923582
- [Background] Banitt M. Evaluation and management of glaucoma after keratoprosthesis. Curr Opin Ophthalmol. 2011 Mar;22(2):133-6. doi: 10.1097/ICU.0b013e328343723d. PMID 21191292
- [Background] Cueva Vargas JL, Belforte N, Di Polo A. The glial cell modulator ibudilast attenuates neuroinflammation and enhances retinal ganglion cell viability in glaucoma through protein kinase A signaling. Neurobiol Dis. 2016 Sep;93:156-71. doi: 10.1016/j.nbd.2016.05.002. Epub 2016 May 6. PMID 27163643
- [Background] Crnej A, Omoto M, Dohlman TH, Dohlman CH, Dana R. Corneal inflammation after miniature keratoprosthesis implantation. Invest Ophthalmol Vis Sci. 2014 Dec 16;56(1):185-9. doi: 10.1167/iovs.14-15884. PMID 25515579
- [Background] Engel LA, Muether PS, Fauser S, Hueber A. The effect of previous surgery and topical eye drops for primary open-angle glaucoma on cytokine expression in aqueous humor. Graefes Arch Clin Exp Ophthalmol. 2014 May;252(5):791-9. doi: 10.1007/s00417-014-2607-5. Epub 2014 Mar 18. PMID 24638257
- [Background] Freedman J, Iserovich P. Pro-inflammatory cytokines in glaucomatous aqueous and encysted Molteno implant blebs and their relationship to pressure. Invest Ophthalmol Vis Sci. 2013 Jul 18;54(7):4851-5. doi: 10.1167/iovs.13-12274. PMID 23788371
- [Background] Burgos-Blasco B, Vidal-Villegas B, Saenz-Frances F, Morales-Fernandez L, Perucho-Gonzalez L, Garcia-Feijoo J, Martinez-de-la-Casa JM. Tear and aqueous humour cytokine profile in primary open-angle glaucoma. Acta Ophthalmol. 2020 Sep;98(6):e768-e772. doi: 10.1111/aos.14374. Epub 2020 Feb 11. PMID 32043817
- [Background] Robert MC, Arafat SN, Spurr-Michaud S, Chodosh J, Dohlman CH, Gipson IK. Tear Matrix Metalloproteinases and Myeloperoxidase Levels in Patients With Boston Keratoprosthesis Type I. Cornea. 2016 Jul;35(7):1008-14. doi: 10.1097/ICO.0000000000000893. PMID 27191670
- [Background] Chen KH, Wu CC, Roy S, Lee SM, Liu JH. Increased interleukin-6 in aqueous humor of neovascular glaucoma. Invest Ophthalmol Vis Sci. 1999 Oct;40(11):2627-32. PMID 10509659
- [Background] Hu DN, Ritch R, Liebmann J, Liu Y, Cheng B, Hu MS. Vascular endothelial growth factor is increased in aqueous humor of glaucomatous eyes. J Glaucoma. 2002 Oct;11(5):406-10. doi: 10.1097/00061198-200210000-00006. PMID 12362079
- [Background] Kuchtey J, Rezaei KA, Jaru-Ampornpan P, Sternberg P Jr, Kuchtey RW. Multiplex cytokine analysis reveals elevated concentration of interleukin-8 in glaucomatous aqueous humor. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6441-7. doi: 10.1167/iovs.10-5216. Epub 2010 Jun 30. PMID 20592224
- [Background] Dohlman CH, Zhou C, Lei F, Cade F, Regatieri CV, Crnej A, Dohlman JG, Shen LQ, Paschalis EI. Glaucoma After Corneal Trauma or Surgery-A Rapid, Inflammatory, IOP-Independent Pathway. Cornea. 2019 Dec;38(12):1589-1594. doi: 10.1097/ICO.0000000000002106. PMID 31453878